CLINICAL TRIAL: NCT02752477
Title: Efficacy of Opioid-free Anesthesia in Reducing Postoperative Pain in Chronic Pain Patients Undergoing Spinal Surgery: A Pilot Study
Brief Title: Efficacy of Opioid-free Anesthesia in Reducing Postoperative Pain in Chronic Pain Patients Undergoing Spinal Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ben Lim (Other)
Responsible Party: Sponsor-Investigator, Ben Lim, Anesthesiologist, University of Saskatchewan
Organization: University of Saskatchewan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO15-253
Record Dates: First submitted 2016-03-29; First posted 2016-04-27 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain; Anesthesia
Keywords: Opioid-sparing
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opioid-free anesthetic (OFA) group (Experimental)
  Interventions: Drug: Opioid-free general anesthetic
- Traditional Anesthesia (TA) group (Active Comparator)
  Interventions: Drug: Traditional general anesthetic

INTERVENTIONS:
Drug: Opioid-free general anesthetic — An opioid-free general anesthetic technique utilizing dexmedetomidine, ketamine, and lidocaine infusions
  Arms: Opioid-free anesthetic (OFA) group
Drug: Traditional general anesthetic — Traditional general anesthetic technique utilizing sufentanil, fentanyl or remifentanil
  Arms: Traditional Anesthesia (TA) group

SUMMARY:
The objective of this trial is to determine whether an opioid-free general anesthetic (OFA) technique utilizing ketamine, dexmedetomidine, and lidocaine infusions can help reduce postoperative pain in opiate-dependent chronic pain patients (CPPs) undergoing spine surgery when compared with traditional opioid-containing techniques. It is expected that this OFA regimen will have a measurable reduction on postoperative opioid consumption and pain scores in CPPs.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain > 6 months, opiate-using patients scheduled for thoracic or lumbar spinal surgery

Exclusion Criteria:

* Pregnant or breastfeeding women, significant hepatic, renal or cardiac disease, allergy to any of the study drugs, inability to consent, respond to pain assessments or use the patient controlled analgesia device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-02 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Quantified opioid-consumption | 48 hours following surgery

SECONDARY OUTCOMES:
Visual analogue scale (VAS) pain scores | 48 hours following surgery
Time of stay in post-anesthetic care unit (PACU) | up to 5 hours following surgery
Incidence of adverse events | 48 hours following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ben Lim, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No